CLINICAL TRIAL: NCT01708642
Title: The Effect of Intraoperative Low Dose Adrenaline on Bleeding in Total Hip Arthroplasty - a Randomized Placebo-controlled Trial
Brief Title: The Effect of Administration of Low Dose Adrenaline During Surgery on Bleeding During Hip Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Oeivind Jans, M.D, Research Fellow, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RH-4074-OJ2; 2012-002889-12 (EudraCT Number)
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Intraoperative Blood Loss
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adrenaline (Experimental): Intraoperative low-dose adrenaline infusion
  Interventions: Drug: Adrenaline
- Placebo (Placebo Comparator): Placebo: Isotonic Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adrenaline — Adrenaline infusion 0.05 microgram / kg / minute
  Other Names: Ephinephrine
  Arms: Adrenaline
Drug: Placebo — Intraoperative isotonic saline infusion as placebo for adrenaline.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of intraoperative administration of low-dose adrenaline on intraoperative blood loss in patients undergoing hip surgery.

DETAILED DESCRIPTION:
Hip arthroplasty is associated with bleeding, anemia and the need for allogeneic transfusion. Administration of low-dose adrenaline activates the coagulation system and may decrease intraoperative and immediate postoperative bleeding. Thus, the aim of this study is to evaluation whether intraoperative IV-administration of low-dose adrenaline reduces bleeding in elective total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Scheduled for primary unilateral hip arthroplasty
* Able to give consent

Exclusion Criteria:

* Allergy towards adrenaline
* Current treatment with: ADP receptor inhibitors or Vitamin K antagonists (within 5 days), Factor Xa inhibitors or Thrombin inhibitors (within 1 day), heparin (excluding low molecular weight heparin for perioperative thromboprophylaxis).
* Current treatment with tricyclic antidepressants
* Use of MAO inhibitors (within previous 14 days) or COMT inhibitors (within 2 days).
* Acute coronary syndrome / myocardial infarction within the previous 6 months.
* not willing to accept blood transfusion
* Participation in other clinical trial within previous 30 days
* Women of childbearing age (without menopause for at least 12 months)
* Glaucoma
* Pheochromocytoma
* Low serum K+ (< 3.0 mmol/L)
* Thyrotoxicosis
* Digoxin intoxication
* Alcohol og drug abuse (investigators judgement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | End of surgery (last suture)
  Intraoperative blood loss as estimated from surgical drain and sponges.

SECONDARY OUTCOMES:
Calculated blood loss | 24 hours after end of surgery.
  Calculated blood loss at 24 h after end of surgery.

OTHER OUTCOMES:
Drug side effects | During surgery (from start of procedure to last suture)
  Side effects causing discontinuation the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Pär I Johanssion, M.D., DMsc., Study Chair — Rigshospitalet, Section for transfusion medicine; Oeivind Jans, M.D., Principal Investigator — Rigshospitalet, Section for Surgical Pathophysiology
Locations (3):
- Denmark (3):
  - Gentofte Hospital, Department of Anaesthesia, Hellerup
  - Hvidovre Hospital, Department of orthopaedic surgery, Hvidovre
  - Vejle Sygehus, Department of orthopedic surgery, Vejle

REFERENCES:
- [Derived] Jans O, Grevstad U, Mandoe H, Kehlet H, Johansson PI. A randomized trial of the effect of low dose epinephrine infusion in addition to tranexamic acid on blood loss during total hip arthroplasty. Br J Anaesth. 2016 Mar;116(3):357-62. doi: 10.1093/bja/aev408. Epub 2016 Jan 27. PMID 26821696